CLINICAL TRIAL: NCT04966195
Title: Stereotactic Body Radiotherapy Based Treatment for Hepatocellular Carcinoma With Extensive Portal Vein Tumor Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: (2016)-050
Record Dates: First submitted 2021-07-11; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2017-06

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Portal Vein Tumor Thrombosis; Stereotactic Body Radiotherapy
Keywords: Hepatocellular carcinoma; Portal vein tumor thrombosis; Stereotactic body radiotherapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: stereotactic body radiotherapy of hepatocellular carcinoma patients with portal vein tumor thrombosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiotherapy (Other): stereotactic body radiotherapy of hepatocellular carcinoma patients with portal vein tumor thrombosis
  Interventions: Radiation: stereotactic body raiotherapy

INTERVENTIONS:
Radiation: stereotactic body raiotherapy — stereotactic body radiotherapy of hepatocellular carcinoma patients with portal vein tumor thrombosis

SUMMARY:
Macrovascular invasion (MVI) is common in HCC, Portal vein tumor thrombus (PVTT) is the most common form of MVI in HCC, with an incidence ranging from 44 to 62.2%. About 10% to 60% of HCC patients have PVTT at the time of diagnosis. the prognosis for those with PVTT remains poor, as their median survival is only 2-4 months via supportive care. There is currently no widely-accepted consensus for the management of HCC with PVTT. According to some guidelines in Europe and America, HCC with PVTT is regarded as Stage C per Barcelona Clinic Liver Cancer (BCLC) Staging system, and sorafenib alone is recommended as the treatment of choice. This study is to analyze the safety and efficacy of radiotherapy of hepatocellular carcinoma patients with portal vein tumor thrombosis.

ELIGIBILITY:
Inclusion Criteria:

1. tumor thrombus involving the main trunk and/or first branches of the portal vein, unsuitable for surgery or TACE;
2. an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2; 3. no refractory ascites;

4. Child-Pugh class A and B, or class C with good performance status; 5. no previous radiotherapy to the liver; 6. more than 700 cc of uninvolved liver

Exclusion Criteria:

1. Have received local or systemic treatments in the past, including but not limited to TACE, immunotherapy, targeted therapy, radiotherapy, radiofrequency therapy, etc.;
2. Diffuse HCC or accompanied by distant metastasis;
3. Severe bleeding tendency or coagulation dysfunction within the previous 6 months;
4. Patients with a history of hepatic encephalopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
overall survival | from enrollment to death (for any reason).assessed up to 12 months
  The time from the patient received treatment to died from any cause

SECONDARY OUTCOMES:
objective response rate | from enrollment to progression or death (for any reason),assessed up to 12 months
  complete or partial response after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- the second affiliated hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No